CLINICAL TRIAL: NCT07096024
Title: Ibrance® Post-Marketing Database Study Incidence of Interstitial Lung Disease in Inoperable or Recurrent Breast Cancer Patients Treated With Palbociclib in a Post-marketing Setting: Cohort Study Using the Medical Data Vision (MDV) Database
Brief Title: A Study to Understand About the Study Medicine Palbociclib in Breast Cancer Patients After it is Out in the Japanese Market
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481117
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Neoplasms
Keywords: Ibrance; Post-Marketing Database Study; Incidence of interstitial lung disease (ILD); inoperable or recurrent breast cancer; palbociclib; Medical Data Vision (MDV)
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Fulvestrant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- New prescription of palbociclib with fulvestrant.: Patients treated with the combination of palbociclib and fulvestrant
  Interventions: Drug: palbociclib plus fulvestrant; Drug: fulvestrant
- New prescription of fulvestrant monotherapy before the launch of palbociclib: Patients treated with fulvestrant alone
  Interventions: Drug: fulvestrant

INTERVENTIONS:
Drug: palbociclib plus fulvestrant — Patients treated with the combination of palbociclib and fulvestrant
  Other Names: Ibrance; fulvestrant
  Groups: New prescription of palbociclib with fulvestrant.
Drug: fulvestrant — Patients treated with fulvestrant alone

SUMMARY:
The purpose of the study is to:

* compare the chances of getting interstitial lung disease (ILD) in new users of palbociclib plus fulvestrant to new users of fulvestrant alone (using data from before palbociclib was out in the market)
* look into the factors that can cause ILD in new users of palbociclib.

This study uses patient data without giving out any personal information of the patient. This data is taken from a hospital-based claims database of the MDV database, that includes data from more than 400 hospitals in Japan.

This study will use data of patients who are:

* diagnosed with breast cancer that include newly treated with palbociclib and/or other endocrine-based therapies for inoperable or recurrent breast cancer between 25 November 2011 and 30 November 2024.

ELIGIBILITY:
Inclusion Criteria:

* Having prescription records of drugs for endocrine therapy (aromatase inhibitors, SERDs, SERMs, and CDK4/6 inhibitors) from 25 November 2011 to 31 December 2024.
* Having any breast cancer records with definitive diagnosis in the same month as the first prescription date.
* Having any records in MDV database on or before 6 months prior to the first prescription date (<= -180 days: first prescription date = 0 day).
* Having any records in MDV database within 6 months prior to the first prescription date (-180 days to 0 day).

Exclusion Criteria:

* Having any records of anti-HER2 medication (e.g., trastuzumab, pertuzumab, lapatinib or trastuzumab emtansine) from 25 November 2011 to 31 December 2024.
* Having any records of second primary cancer with definitive diagnosis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The source population comprises patients diagnosed with breast cancer that include newly treated with palbociclib and/or other endocrine-based therapies for inoperable or recurrent breast cancer between 25 November 2011 and 31 December 2024
Sampling Method: Probability Sample
Enrollment: 1772 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-02-07 (Actual); Study Completion 2025-02-07 (Actual)

PRIMARY OUTCOMES:
The hazard ratios of ILD in palbociclib plus fulvestrant to new users of fulvestrant alone | 25 November 2011 and 30 September 2024
The rate ratios of ILD in palbociclib plus fulvestrant to new users of fulvestrant alone | 25 November 2011 and 30 September 2024
The rate differences of ILD in palbociclib plus fulvestrant to new users of fulvestrant alone | 25 November 2011 and 30 September 2024
The incidence rate of ILD by each risk factor in new users of palbociclib | 25 November 2011 and 30 September 2024

SECONDARY OUTCOMES:
The incidence rate of ILD by each risk factor in new users of endocrine-based therapies including combination with CDK4/6 inhibitors | 25 November 2011 and 30 September 2024

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New York, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.